CLINICAL TRIAL: NCT00143676
Title: A Double-blind, Randomized Placebo-controlled Study to Evaluate the Efficacy and Safety of TAK-475 50 mg, 100 mg, or Placebo When Co-administered With Atorvastatin (10 mg to 40 mg) in Subjects With Primary Hypercholesterolemia
Brief Title: Efficacy of Lapaquistat Acetate and Atorvastatin on Blood Cholesterol Levels in Subjects With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-475-009; U1111-1122-7783 (Registry Identifier: WHO)
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lapaquistat Acetate 50 mg QD + Atorvastatin (Experimental)
  Interventions: Drug: Lapaquistat acetate and atorvastatin
- Lapaquistat Acetate 100 mg QD + Atorvastatin (Experimental)
  Interventions: Drug: Lapaquistat acetate and atorvastatin
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Lapaquistat acetate and atorvastatin — Lapaquistat acetate 50 mg, tablets, orally, once daily and Atorvastatin 10 mg to 40 mg stable dose for up to 24 weeks.
  Other Names: Lapaquistat; Lipitor; TAK-475
  Arms: Lapaquistat Acetate 50 mg QD + Atorvastatin
Drug: Lapaquistat acetate and atorvastatin — Lapaquistat acetate 100 mg, tablets, orally, once daily and Atorvastatin 10 mg to 40 mg stable dose for up to 24 weeks.
  Other Names: Lapaquistat; Lipitor; TAK475
  Arms: Lapaquistat Acetate 100 mg QD + Atorvastatin
Drug: Atorvastatin — Lapaquistat acetate placebo-matching tablets, orally, once daily and Atorvastatin 10 mg to 40 mg stable dose for up to 24 weeks.
  Other Names: Lipitor
  Arms: Atorvastatin

SUMMARY:
The purpose of this study is to determine the efficacy of lapaquistat acetate, once daily (QD), on lowering cholesterol in subjects already taking atorvastatin.

DETAILED DESCRIPTION:
According to the World Health Organization, CHD is now the leading cause of death worldwide. In 2001, CHD caused 7.2 million deaths and estimates for 2020 indicate that annual CHD deaths will increase to 11.1 million. These statistics suggest that improved options are needed to treat hypercholesterolemia and dyslipidemia.

The balance among cholesterol synthesis, dietary intake, and degradation is normally adequate to maintain healthy cholesterol plasma levels. However, in patients with hypercholesterolemia, elevated low-density lipoprotein cholesterol leads to atherosclerotic deposition of cholesterol in the arterial walls. Consequently, in this population it has been established that lowering low-density lipoprotein cholesterol plasma concentrations effectively reduces cardiovascular morbidity and mortality. The National Cholesterol Education Program Adult Treatment Panel III has therefore identified control of low-density lipoprotein cholesterol as essential in the prevention and management of CHD. Additional lipid risk factors designated by National Cholesterol Education Program Adult Treatment Panel III include elevated triglycerides, elevated non-high-density lipoprotein cholesterol (atherogenic lipoproteins), and low levels of high-density lipoprotein cholesterol. Lipoproteins rich in triglycerides, such as very-low-density lipoprotein cholesterol, appear to contribute to atherosclerosis, whereas the apparent protective effect of high-density lipoprotein cholesterol, which is likely related to high-density lipoprotein cholesterol-facilitated transport of cholesterol away from atherosclerotic deposits, may be limited at low high-density lipoprotein cholesterol concentrations.

Initial dietary and lifestyle measures taken to control dyslipidemia are often inadequate, and most patients require pharmacologic intervention. Currently, 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors (statins) are the first-line monotherapies most often prescribed to reduce low-density lipoprotein cholesterol, after diet and therapeutic lifestyle change. However, with statin monotherapy, many patients fail to reach National Cholesterol Education Program Adult Treatment Panel III recommended levels of low-density lipoprotein cholesterol reduction. As a result, the statin dosage must be increased or an additional treatment added to achieve treatment goals. Increasing the statin dosage may result in decreased tolerability and potential safety concerns, contributing to the high discontinuation rates of statins and their prescription at low and often ineffective doses. Further, although the effectiveness of increasing the dose varies among the statins, in general, doubling of the dose above the minimum effective dose has been found to decrease serum low-density lipoprotein cholesterol by only an additional 6 percent.

TGRD is developing an orally active squalene synthase inhibitor, TAK-475 (lapaquistat acetate) for the treatment of dyslipidemia. Lapaquistat acetate inhibits the biosynthesis of cholesterol by inhibiting the enzyme squalene synthase, which catalyzes the conversion of farnesyl diphosphate to squalene-a precursor in the final steps of cholesterol production.

This study will assess the effects of co-administration of lapaquistat acetate with atorvastatin, the most commonly prescribed statin in the United States, on LDL-C and associated lipid variables in subjects with hypercholesterolemia. Study Participation is anticipated to be up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of childbearing potential must not be pregnant as determined by a negative serum human chorionic gonadotropin, lactating, or planning on becoming pregnant, and agrees to use acceptable forms of contraception during the study.
* Must have a mean low density lipoprotein cholesterol value greater than or equal to 2.590 mmol/L (100 mg/dL) for 2 consecutive samples
* Must have a mean triglyceride value less than or equal to 4.516 mmol/L (400 mg/dL) for 2 consecutive samples.
* Has taken a stable dose of atorvastatin (10 to 40 mg)
* Has clinical laboratory evaluations within reference range for the testing laboratory.
* Is willing and able to continue to comply with a standardized low-cholesterol diet.

Exclusion Criteria:

* Has an alanine aminotransferase or aspartate aminotransferase level greater than 1.5 times the upper limit of normal, active liver disease or jaundice.
* Has a serum creatinine level greater than 135 μmol/L (1.5 mg/dL).
* Has a creatine phosphokinase level greater than 3 times the upper limit of normal
* Has diabetes with a hemoglobin A1c level greater than 8% at Visit 1.
* Has a history of cancer in remission for less than 5 years prior to the first dose of study drug.
* Has an endocrine disorder, such as Cushing's syndrome, hyperthyroidism, or inappropriately treated hypothyroidism, affecting lipid metabolism.
* Has a history of myocardial infarction, unstable angina, transient ischemic attacks, cerebrovascular accident, percutaneous coronary intervention, or coronary or peripheral arterial surgery.
* Has a positive hepatitis B surface antigen, or hepatitis C virus antibody, as determined by medical history and/or the subject's verbal report.
* Has a positive human immunodeficiency virus status or was taking antiretroviral medications as determined by medical history and/or the subject's verbal report.
* Has had exposure to lapaquistat acetate in other studies, was participating in another investigational study, or had participated in an investigational study within the past 30 days or, for drugs with a long half-life, within a period of less than 5 times the drug's half-life.
* Has a known hypersensitivity or history of adverse reaction to atorvastatin.
* Has a history or presence of clinically significant food allergy that would prevent adherence to the recommended diet.
* Has a known homozygous familial hypercholesterolemia or known type III hyperlipoproteinemia.
* Has fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain.
* Has uncontrolled hypertension
* Has inflammatory bowel disease or any other malabsorption syndrome or has had gastric bypass or any other surgical procedure for weight loss.
* Has a history of drug abuse or a history of alcohol abuse within the past 2 years.
* Has any other serious disease or condition that might reduce life expectancy, impair successful management according to the protocol, or make the subject an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2005-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Low Density Lipoprotein cholesterol | Week 24 or Final Visit

SECONDARY OUTCOMES:
Adverse Events | Weeks: 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Physical Examination | Week 24 or Final Visit
Safety Laboratory Tests | Weeks: 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Electrocardiogram assessments | Week 24 or Final Visit
Best Corrected Visual Acuity results | Week 24 or Final Visit
Vital Signs | Weeks: 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Change from Baseline in Triglycerides | Week 24 or Final Visit
Change from Baseline in Total Cholesterol | Week 24 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in Very Low Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in apolipoprotein A1 | Week 24 or Final Visit
Change from Baseline in apolipoprotein B | Week 24 or Final Visit
Change from Baseline in non- High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of Low Density Lipoprotein cholesterol/High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of Total Cholesterol/High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of apolipoprotein A1/apolipoprotein B | Week 24 or Final Visit
Change from Baseline in high-sensitivity C-reactive protein | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 1.813 mmol/L (70 mg/dL) | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 2.590 mmol/L (100 mg/dL) | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 3.367 mmol/L (130 mg/dL) | Week 24 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (78):
- United States (78):
  - Birmingham, Alabama
  - Northport, Alabama
  - Sierra Vista, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Searcy, Arkansas
  - Anaheim, California
  - Carmichael, California
  - Chula Vista, California
  - Escondido, California
  - Pismo Beach, California
  - Santa Rosa, California
  - Golden, Colorado
  - Waterbury, Connecticut
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - West Palm Beach, Florida
  - Honolulu, Hawaii
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Peoria, Illinois
  - Bloomington, Indiana
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Waterloo, Iowa
  - Arkansas City, Kansas
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Auburn, Maine
  - Livonia, Michigan
  - Edina, Minnesota
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Edison, New Jersey
  - Margate City, New Jersey
  - New Hyde Park, New York
  - Rochester, New York
  - Syracuse, New York
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Altoona, Pennsylvania
  - Downingtown, Pennsylvania
  - Sellerville, Pennsylvania
  - Tipton, Pennsylvania
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Chattanooga, Tennessee
  - Morristown, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Euless, Texas
  - San Antonio, Texas
  - The Colony, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Renton, Washington
  - Madison, Wisconsin

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985